CLINICAL TRIAL: NCT06759168
Title: Impact of Cataract Surgery on the Incidence and Progression of Dry Eye Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Nabil Habeb, resident doctor, Assiut University
Other Study IDs: Dry eye & cataract surgery
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Dry Eye
Keywords: Dry eye; Cataract surgery
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Relation between dry eye and cataract

DETAILED DESCRIPTION:
Study the impact of cataract surgery on the incidence and progression of dry eye disease

ELIGIBILITY:
Inclusion Criteria:

* patients aged above 40-years old undergoing cataract surgery
* patients without dry eye disease
* patients with mild to moderate degree of dry eye disease Both gender, male and female

Exclusion Criteria:

* patients aged less 40-year old undergoing cataract surgery
* patients with severe degrees of dry eye disease
* patients with autoimmune disease
* patients with chronic blepharitis

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Both males and females above 40- year old going cataract surgery
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Dry eye after cataract surgery | 1 week, 1 month and 3 months
  The incidence of new or working dry eye symptoms following cataract surgery

SECONDARY OUTCOMES:
risk factors to dry eye | 1 month
  Identification of risk factors associated with postoperative dry eye

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ram J, Gupta A, Brar G, Kaushik S, Gupta A. Outcomes of phacoemulsification in patients with dry eye. J Cataract Refract Surg. 2002 Aug;28(8):1386-9. doi: 10.1016/s0886-3350(02)01387-1. PMID 12160808
- [Background] Shaaban YM, Aziz BF. Tear film assessment before and after phacoemulsification in patients with age-related cataracts. BMC Ophthalmol. 2024 Jul 11;24(1):280. doi: 10.1186/s12886-024-03542-2. PMID 38992580